CLINICAL TRIAL: NCT01185652
Title: A Study on Smoking-related Lung Function Abnormalities and Correlation With Serum Biomarkers in Chinese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: David Chi-leung LAM, University of Hong Kong
Other Study IDs: HKCTR803
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Airflow Obstruction
Keywords: Smoking; airflow obstruction; pulmonary function tests
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml Peripheral blood will be collected upon recruitment for storage and later extraction of DNA and serum biomarkers
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Tobacco-smoking causes lung function decline with airflow obstruction, which may be accelerated in persistent smokers.This would eventually lead to chronic obstructive pulmonary disease (COPD), a leading cause of morbidity and mortality in Hong Kong and globally. Lung function decline is gradual and not appreciated by the smoker until damage is advanced, and often under-recognised in the early stages of disease by healthcare providers. Spirometry is an established lung function measurement tool, and the most simple objective method to detect lung function decline. There is literature suggesting that newer spirometric parameters, FEV3 and FEV6, which are easier to achieve in the measurement process than conventional parameters, are comparable alternatives in detecting lung function decline.

The aims of this study are:

1. to evaluate and compare lung function decline in persistent smokers and non-smokers
2. to study the usefulness of FEV3/FVC and FEV1/FEV6 in detecting lung function decline
3. to correlate symptom scores with lung function parameters
4. To correlate serum biomarker levels with respiratory symptoms and lung function parameters in smokers and non-smokers

This is a follow-up study on a territory wide cohort including smokers and non-smokers, who have undergone lung function testing in 2001-03. Subjects will be invited to have repeat lung function assessment.

The hypotheses of this study are:

1. smokers have significantly greater decline in lung function compared to non-smokers in Hong Kong Chinese;
2. newer lung function parameters are useful alternatives in detecting lung function decline
3. serum inflammatory biomarker (IL-8, TGF-β, MMP9, TIMP-1, CRP) levels correlate with respiratory symptoms and lung function parameters in smokers when compared with non-smokers

DETAILED DESCRIPTION:
Tobacco-smoking causes lung function decline with airflow obstruction, which may be accelerated in persistent smokers.This would eventually lead to chronic obstructive pulmonary disease (COPD), a leading cause of morbidity and mortality in Hong Kong and globally. Lung function decline is gradual and not appreciated by the smoker until damage is advanced, and often under-recognised in the early stages of disease by healthcare providers. Spirometry is an established lung function measurement tool, and the most simple objective method to detect lung function decline. There is literature suggesting that newer spirometric parameters, FEV3 and FEV6, which are easier to achieve in the measurement process than conventional parameters, are comparable alternatives in detecting lung function decline.

The aims of this study are:

1. to evaluate and compare lung function decline in persistent smokers and non-smokers
2. to study the usefulness of FEV3/FVC and FEV1/FEV6 in detecting lung function decline
3. to correlate symptom scores with lung function parameters
4. To correlate serum biomarker levels with respiratory symptoms and lung function parameters in smokers and non-smokers

This is a follow-up study on a territory wide cohort including smokers and non-smokers, who have undergone lung function testing in 2001-03. Subjects will be invited to have repeat lung function assessment.

The demonstration of excessive lung function decline in the local smoking population would reinforce the anti-tobacco message in the community. Establishing the practical utility of newer lung function parameters can help to disseminate their utilization for early objective health information, which would provide incentives for healthcare professionals as well as individual smokers in the pursuance of smoking cessation.

The hypotheses of this study are:

1. smokers have significantly greater decline in lung function compared to non-smokers in Hong Kong Chinese;
2. newer lung function parameters are useful alternatives in detecting lung function decline
3. serum inflammatory biomarker (IL-8, TGF-β, MMP9, TIMP-1, CRP) levels correlate with respiratory symptoms and lung function parameters in smokers when compared with non-smokers

Subjects In 2001 - 2003, we conducted a multi-center study to recruit 1089 non-smokers for establishing local reference lung function values, and 694 smokers for investigating the diagnostic definition of airflow obstruction. The cohort was derived from a random population sample and the characteristics of the two cohorts have been described in detail in previous communications. All subjects will be invited to return for spirometry testing. We would compare their lung function parameters 7 years ago with the repeat measurements obtained in this study.

Methods:

i. Subjects will be interviewed using a questionnaire based on the ATS Questionnaire for Chronic Respiratory Symptoms. In addition, a detailed smoking history will be asked; for those who have given up smoking in the interval between the previous study and this study, the time of quitting will be recorded.

ii. Spirometry. Spirometry with bronchodilator testing will be performed according to the ATS-ERS guidelines, using Sensormedics Vmax 229. All participating centers are experienced in lung function testing. Quality control of the tests will be ensured by 1) standardization and calibration of the equipments prior to commencement of study, 2) briefing session for all involved technicians conducted by a senior technician, 3) technical quality of raw data will be scrutinized by a respiratory specialist iii. Seum biomarkers Recruited subjects will be invited to give 10 ml blood in the same lung function test session.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Agreed to give informed written consent

Exclusion Criteria:

* subjects refuse to give informed written consent
* subjects with active infection or medical illness under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 2001 - 2003, we conducted a study to recruit 1089 non-smokers for establishing local reference lung function values, and 694 smokers for investigating the diagnostic definition of airflow obstruction. The cohort was derived from a random population sample and the characteristics of the two cohorts have been described in detail in previous communications. All subjects will be invited to return for spirometry testing (at one of the participating hospitals of their choice) and an interview. We would compare their lung function parameters 7 years ago with the repeat measurements obtained in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-04 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Spirometry parameters | Two years
  1. FEV1 raw,
  2. FEV1 % predicted
  3. FEV1/FVC
  4. FEV3 raw
  5. FEV3/FVC
  6. FEV1/FEV6

SECONDARY OUTCOMES:
Serum biomarkers | Two years
  Serum levels of IL-8, TGF-β, MMP9, TIMP-1, CRP

CONTACTS AND LOCATIONS:
Overall Officials: David CL Lam, BSc,MBBS,PhD,FCCP,FACP,FRCP(E), Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lam DC, Kwok HH, Yu WC, Ko FW, Tam CY, Lau AC, Fong DY, Ip MS. CC16 levels correlate with cigarette smoke exposure in bronchial epithelial cells and with lung function decline in smokers. BMC Pulm Med. 2018 Mar 16;18(1):47. doi: 10.1186/s12890-018-0607-7. PMID 29548305